CLINICAL TRIAL: NCT00937716
Title: Treatment Response in Schizophrenia: Bridging Imaging and Postmortem Studies
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Adrianne C Lahti, Professor & Division Director of Behavioral Neurobiology, University of Alabama at Birmingham
Other Study IDs: F080807011
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; treatment response; risperidone; functional magnetic resonance; functional magnetic spectroscopy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be tested for dopamine, serotonin, norepinephrine, and glutamine-related genes. In previous studies, all of these neurotransmitters have been associated with schizophrenia and/or schizoaffective disorder.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diagnosis of Schizophrenia: Patients with a diagnosis of schizophrenia that have been off antipsychotic medicine and would like to resume treatment will be enrolled in the study.
- Healthy Volunteers: Healthy Volunteers without a psychiatric diagnosis, central nervous system condition, serious head injury, or current drug use will be matched on an individual basis to schizophrenic participants and used as a control population.

SUMMARY:
The overarching goal is to identify imaging markers that will predict treatment response, and to confirm or validate these biomarkers using anatomical studies of postmortem tissue. Early detection of drug response would yield specific treatment strategies that are tailored to the individual, thus improving both the quality of life of the patients and drastically reducing the costs associated with unsuccessful treatment strategies.

DETAILED DESCRIPTION:
Our past brain imaging and Positron Emission Tomography (PET) studies have contributed to the understanding of specific brain regions related to treatment response to antipsychotic drugs in schizophrenia. We have found that treatment response to antipsychotic medication is related to blood-flow patterns in specific regions (such as the ventral striatum, anterior cingulate cortex, and hippocampus). In addition, functional changes in these regions following one week of antipsychotic drug therapy are predictive of treatment response. Dr. Roberts, a neuroanatomist, has studied the post mortem (after death) brains of patients with schizophrenia while working in association with the Maryland Brain Collection. Her studies have indicated an increased number of dopaminergic synapses (that is, neurons that produce the neurotransmitter dopamine) in these regions in patients who were known to have had a favorable response to antipsychotic drug therapy. In addition, from this post-mortem work we know the number of glutamate synapses in these regions were significantly different between good treatment responders and poor responders.

From these studies we have hypothesized that in schizophrenia an over-abundance of dopamine in the ventral striatum interferes with normal functioning by limiting the transmission of glutamate. Putatively, antipsychotic medications may decrease the symptoms of schizophrenia by restoring glutamatergic activity in the ventral striatum and projected areas, such as the anterior cingulate cortex and hippocampus. We have hypothesized that those individuals responding favorably to antipsychotic drug therapy will display greater glutamate activity in the ventral striatum (due to dopamine blockade) and the other regions receiving glutamate projections. This should lead to restored neuronal functioning in good responders when compared to treatment resistant and poor responders to antipsychotic drug treatment. We will test this hypothesis using complementary imaging and postmortem studies yielding data that will permit the formulation of a comprehensive model for antipsychotic drug responses in subjects with severe mental illness.

Magnetic Resonance is a technique for probing atoms and molecules based upon their interaction with an external magnetic field. Magnetic Resonance does not use ionizing radiation. The most familiar example of this is Magnetic Resonance Imaging (MRI). Another application of Magnetic Resonance is called functional Magnetic Resonance Imaging (fMRI). Functional Magnetic Resonance Imaging (fMRI) allows us to measure the Blood Oxygenation Level-Dependent (BOLD) response, a measure of blood flow in the brain that is known to correlate with neuronal activity. Another application of Magnetic Resonance is Magnetic Resonance Spectroscopy (MRS), which allows the measurements of specific metabolites such as N-acetyl aspartate (NAA), a measure of neuronal integrity, and Glutamate, which is involved in neurotransmission and metabolism. We will seek to replicate and extend our past Positron Emission Tomography (PET) findings with functional magnetic resonance imaging (fMRI) using cognitive tasks that are known to activate the hippocampus (Episodic memory task) and the anterior cingulate cortex (Stroop task). This aim will further seek to parse out the differential contribution of the hippocampus and the anterior cingulate cortex to treatment response. At the same time, N-acetylaspartate, a marker of neuronal integrity, and glutamate measurements obtained with magnetic resonance spectroscopy in the anterior cingulate cortex and hippocampus will directly probe in the living brain the relation between neuronal integrity, glutamate function, and treatment response. In parallel, the postmortem work of Dr. Roberts (UAB IRB exemption: NO70813001, IRB#F080306003) will concentrate on the study of the anterior cingulate cortex in post mortem brains of schizophrenic patients. These studies should allow the development of hypotheses about the pathophysiology of treatment response and provide a basis for the interpretation of functional imaging data. The overarching goal is to identify imaging markers that will predict treatment response, and to confirm or validate these biomarkers using anatomical studies of postmortem tissue. Early detection of drug response would yield specific treatment strategies that are tailored to the individual, thus improving both the quality of life of the patients and drastically reducing the costs associated with unsuccessful treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers or schizophrenic patients between the age of 19 and 55.

Exclusion Criteria:

* Individuals with a diagnosable central nervous system illness.
* Major medical condition, active substance abuse or dependence, pregnancy, or history of head trauma.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit fifty patients with a diagnosis of schizophrenia presenting at UAB clinics who have stopped taking APD medication for at least 10 days and agree to antipsychotic treatment, and twenty-five matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate whether MRI signals (both fMRI and 1H-MRS) predictive of treatment response to antipsychotic therapy in schizophrenia. | at conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne C Lahti, MD, Principal Investigator — University of Alabama at Birmingham, Department of Psychiatry
Locations (1):
- University of Alabama at Birmingham, Department of Psychiatry, SC 501, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No